CLINICAL TRIAL: NCT05279742
Title: Enhancing the Natriuretic Peptide System in HFpEF: A Randomized Double-Blind Placebo-Controlled Triple Crossover Study
Brief Title: Enhancing the Natriuretic Peptide System in HFpEF
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Horng Chen (Other)
Responsible Party: Sponsor-Investigator, Horng Chen, Regulatory Sponsor, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 21-008978
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Chronic Kidney Diseases
Keywords: Exercise Induced Dyspnea
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- HFpEF-CKD with MANP and oral placebo (Experimental): Subjects with with HFpEF volume overload in the presence of chronic kidney diseases and clinical symptoms at rest (e.g. peripheral edema, weight gain, and abdominal distention) will receive study drug MANP and an oral placebo followed by a 1 week washout period.
  Interventions: Drug: MANP; Drug: Oral Placebo
- HFpEF-EI with MANP and oral placebo (Experimental): Subjects with with HFpEF with exercise induced dyspnea (difficult or labored breathing) without clinical symptoms at rest (e.g. peripheral edema, weight gain, and abdominal distention) will receive study drug MANP and an oral placebo followed by a 1 week washout period.
  Interventions: Drug: MANP; Drug: Oral Placebo
- HFpEF-CKD with Sacbitril/Valsartan with an injected placebo (Experimental): Subjects with with HFpEF volume overload in the presence of chronic kidney diseases and clinical symptoms at rest (e.g. peripheral edema, weight gain, and abdominal distention) will receive study drug Sacbitril/Valsartan and an injected placebo followed by a 1 week washout period.
  Interventions: Drug: Sacubitril/Valsartan; Drug: Injection Placebo
- HFpEF-EI with Sacbitril/Valsartan with an injected placebo (Experimental): Subjects with with HFpEF with exercise induced dyspnea (difficult or labored breathing) without clinical symptoms at rest (e.g. peripheral edema, weight gain, and abdominal distention) will receive study drug Sacbitril/Valsartan and an injected placebo followed by a 1 week washout period.
  Interventions: Drug: Sacubitril/Valsartan; Drug: Injection Placebo
- HFpEF-CKD with an oral and injected placebo (Placebo Comparator): Subjects with with HFpEF volume overload in the presence of chronic kidney diseases and clinical symptoms at rest (e.g. peripheral edema, weight gain, and abdominal distention) will receive an oral and injected placebo followed by a 1 week washout period.
  Interventions: Drug: Oral Placebo; Drug: Injection Placebo
- HFpEF-EI with an oral and injected placebo (Placebo Comparator): Subjects with with HFpEF with exercise induced dyspnea (difficult or labored breathing) without clinical symptoms at rest (e.g. peripheral edema, weight gain, and abdominal distention) will receive an oral and injected placebo followed by a 1 week washout period.
  Interventions: Drug: Oral Placebo; Drug: Injection Placebo

INTERVENTIONS:
Drug: MANP — Single subcutaneous injection 5 µg/Kg
  Arms: HFpEF-CKD with MANP and oral placebo; HFpEF-EI with MANP and oral placebo
Drug: Sacubitril/Valsartan — Oral single dose 97/103 mg
  Other Names: Entresto
  Arms: HFpEF-CKD with Sacbitril/Valsartan with an injected placebo; HFpEF-EI with Sacbitril/Valsartan with an injected placebo
Drug: Oral Placebo — Oral single dose that contains no active ingredient
  Arms: HFpEF-CKD with MANP and oral placebo; HFpEF-CKD with an oral and injected placebo; HFpEF-EI with MANP and oral placebo; HFpEF-EI with an oral and injected placebo
Drug: Injection Placebo — Single subcutaneous injection that contains no active ingredient
  Arms: HFpEF-CKD with Sacbitril/Valsartan with an injected placebo; HFpEF-CKD with an oral and injected placebo; HFpEF-EI with Sacbitril/Valsartan with an injected placebo; HFpEF-EI with an oral and injected placebo

SUMMARY:
The purpose of this study is to look at the differences in how individuals with heart failure with preserved ejection fraction in the presence of chronic kidney disease (HFpEF-CKD) and exercise induced dyspnea without objective findings of fluid retention (HFpEF-EI) bodies function using drugs Sacubatril/Valsartan (Entresto) and MANP.

DETAILED DESCRIPTION:
Visit 1

Consent Visit: Possible study participants will meet with study coordinator to review consent form. After enrollment into the study. Diet instructions will be given by a dietician about a no added salt diet, 120 mEq Na/day, which will be maintained throughout the study period. Comprehensive metabolic panel and complete blood count with differential and uring pregnancy test (for premenopausal women) will be obtained as well as a brief physical exam or nursing assessment. Visit 2 will be scheduled at least one week out from consent visit to accommodate diet compliance, unless participant is already compliant with salt intake parameter. Instructions for completing a 24-hour urine collection, and container for Study Visit 2, will be given.

Subjects who are taking angiotensin converting enzyme inhibitors (ACEI) will be switched over to an equivalent dose of Valsartan or Losartan which will be maintained for the rest of the study period.

Visit 2

Participants will start a twenty-four hour urine collection one day prior to the active study day.

Subjects will be admitted to the CRU. First urine void after admission collected (Visit 2 Study Day only). A physical exam or nursing assessment will be done as well as a urine pregnancy test (for premenopausal women). On the active study day, subjects will withhold their usual dose of medications and will be placed in the supine position for 1 hour. During the first 15 minutes, two standard intravenous (IV) catheters will be placed (one in each arm). One catheter will be used for infusion and the other (in the contralateral arm) for blood sampling. A bladder ultrasound will be completed after the participant's first void after admitting to assess for urine retention. Subjects will be asked to drink 10ml/Kg of water to insure sufficient urinary flow. A priming dose (calculated according to body size) of Iohexol, to measure glomerular filtration rate (GFR), is infused, followed by a constant rate IV sustaining dose (calculated according to estimated kidney function) of Iohexol. The subjects will be asked to empty their bladder spontaneously every thirty minutes (if subjects are unable to void every thirty minutes, a urinary catheter will be used upon consent). Throughout the study, at the end of each 30-minute clearance period, subjects will be asked to drink an amount of water equivalent to the sum of the blood losses and the urinary flow.

Blood pressure will be measured at 20-minute intervals by using an automatic blood pressure cuff, and heart rate will be continuously monitored by electrocardiography. Echocardiography will be performed during these baseline clearances to determine left atrial (LA) and LV volumes and systolic and diastolic function.

After the baseline clearance, the subjects will be randomized to receive either a) double placebo (oral and SQ) or b) Oral Sacubatril/valsartan (Entresto 97/103 mg) + SQ placebo or c) SQ MANP (5 µg/Kg) + oral placebo. One hour after the administration of the oral medication, the SQ injection will be administered. Thirty minutes after the administration of SQ injection, the acute saline load will be administered (normal saline 0.9% 0.25 ml/kg/min for 1 hour). Two 30-minute clearances (as outlined above) will be repeated with the subjects in a supine position during the saline infusion. As above, blood samples are collected midway during each clearance and urine samples are obtained every 30 minutes. Echocardiography will be repeated immediately after the end of the saline infusion, after which subjects will be allowed to eat a meal and be dismissed.

The subjects will return after at least 1 week of washout for the second crossover study

Visit 3

Visit 3 will take place the same as described in Visit 2, receiving one of the 2 medication administrations not received on Visit 2: (a) double placebo (oral and SQ) or b) Oral Sacubatril/valsartan (Entresto 97/103 mg) + SQ placebo or c) SQ MANP (5 µg/Kg) + oral placebo).

The subjects will return again after at least 1 week of washout for the third crossover study.

Visit 4

Visit 4 will take place the same as described in Visit 2, receiving the remaining of the medication administrations not received on Visit 2 or Visit 3: (a) double placebo (oral and SQ) or b) Ora Sacubatril/valsartan (Entresto 97/103 mg) + SQ placebo or c) SQ MANP (5 µg/Kg) + oral placebo).

At the end of Visit 4, study participation is complete.

ELIGIBILITY:
Inclusion Criteria:

Group 1: HFpEF-CKD-will consist of 30 subjects with:

* Ejection fraction of equal or greater than 55%; and
* Evidence of increased LV filling pressures, including at least 2 of the following: average septal-lateral E/e' ratio ≥ 15; tricuspid regurgitation (TR) peak velocity > 2:8 m/s;
* Left atrial volume index >34mL/m^2 assessed by echocardiography; and
* Previous diagnosis of HF with New York Heart Association (NYHA) functional class II-III symptoms on chronic diuretic therapy; and
* CKD defined as glomerular filtration rate (eGFR) of 15-80 mL/min/1.73 m^2 as estimated by the Modification of Diet in Renal Disease equation. Subject needs to be on stable dose of chronic diuretic for at least 4 weeks prior to study and maintained on the same dose for the duration of the study. In addition to the exclusion criteria listed below, to ensure a more homogenous group of subjects, we will exclude subjects with Diabetes or BMI > 35 (because endogenous natriuretic peptide levels are low in obese subjects).

Group 2: HFpEF-EI-will consist of 30 subjects with:

* Ejection fraction of equal or greater than 55%; and
* Previous invasive determination of normal pulmonary capillary wedge pressure ≤ 15 mmHg) at rest and ≥ 25 mmHg during exercise; and
* New York Heart Association (NYHA) functional class II-III symptoms; and
* Glomerular filtration rate (eGFR) of > 50 mL/min/1.73 m^2 as estimated by the Modification of Diet in Renal Disease equation. In addition to the exclusion criteria listed below, to ensure a more homogenous group of subjects, we will exclude subjects with Diabetes or BMI>35 (because endogenous natriuretic peptide levels are low in obese subjects).

Exclusion Criteria:

* Body mass index > 35.
* Blood pressure < 100/60 or > 180/100 mmHg.
* Diabetes.
* Myocardial infarction within 6 months of screening.
* Unstable angina within 6 months of screening, or any evidence of myocardial ischemia.
* Significant valvular heart diseases.
* Hypertrophic, restrictive or obstructive cardiomyopathy.
* Constrictive pericarditis.
* Primary pulmonary hypertension.
* Biopsy proven active myocarditis.
* Severe congenital heart diseases.
* Cardiac amyloidosis.
* Fabry disease.
* Sarcoidosis.
* Sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening.
* Second or third degree heart block without a permanent cardiac pacemaker.
* Stroke within 3 months of screening, or other evidence of significantly compromised CNS perfusion.
* Hemoglobin < 9 g/dl
* ALT > 2 times the upper limit of normal;
* Serum sodium of < 135 mEq/dL or > 150 mEq/dL
* Serum potassium of < 3.5 mEq/dL or > 5.7 mEq/dL.
* Other acute or chronic medical conditions or laboratory abnormality which may increase the risks associated with study participation or may interfere with interpretation of the data.
* Received an investigational drug within 1 month prior to dosing.
* Patients with an allergy to iodine;
* female subject who is pregnant or breastfeeding.
* In the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in Plasma ANP | 24 hours
  Change in Plasma ANP (pg/ml) level after administration of study drug/placebo compared to baseline in response to volume expansion in HFpEF-EI vs HFpEF-CKD.
Change in Composite Score of cGMP, sodium excretion, GFR, and Anx-A1 Plasma cGMP, urinary cGMP, urinary sodium excretion, GFR, ANX-A1acute VE with MANP | 24 hours
  A composite score of change in urinary cGMP (pmol/min), sodium excretion (mEq/min), GFR (ml/min), and Anx-A1 (pg/ml) after administration of study drug/placebo compared to baseline in response to volume expansion in HFpEF-EI vs HFpEF-CKD within each treatment group.

SECONDARY OUTCOMES:
Change in Plasma NT-pro BNP | 24 hours
  Change in Plasma NT-pro BNP (pg/ml) after administration of study drug/placebo compared to baseline in response to volume expansion in HFpEF-EI vs HFpEF-CKD.
Change in Plasma cGMP | 24 hours
  Change in plasma cGMP (pmol/ml) after administration of study drug/placebo compared to baseline in response to volume expansion in HFpEF-EI vs HFpEF-CKD.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M McKie, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No